CLINICAL TRIAL: NCT02128607
Title: Immediate and Short-term Effects of Mulligan "Sustained Natural Apophyseal Glides" for a Subgroup of Low Back Pain Patients: A Randomized Placebo Controlled Trial
Brief Title: A Randomized Placebo Controlled Trial on the Efficacy of Sustained Natural Apophyseal Glide (SNAG) in Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Benjamin Hidalgo, PhD-s, assistant-teacher, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IoNS-UCL-Hidalgo-02
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Low Back Pain; Manual Therapy; Sustained Natural Apophyseal Glide (SNAG)
Keywords: low back pain; manual therapy; Mulligan; sustained natural apophyseal glide (SNAG); Kinematic spine model
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real SNAG (Active Comparator): A real sustained natural apophyseal glide (SNAG / Mulligan technique) applied on the lumbar spine from a sitting position, and in a trunk flexion direction with the use of the belt.
  Interventions: Device: SNAG
- Sham SNAG (Placebo Comparator): A sham (placebo) sustained natural apophyseal glide (SNAG / Mulligan technique) applied on the lumbar spine from a sitting position, and in a trunk flexion direction with the use of the belt.
  Interventions: Device: Sham

INTERVENTIONS:
Device: SNAG — sustained natural apophyseal glide: SNAG / Mulligan technique
  Arms: Real SNAG
Device: Sham
  Arms: Sham SNAG

SUMMARY:
Objectives:

Determine the efficacy of the SNAG technique (Mulligan) applied to a subgroup of people with non-specific low back pain (LBP) on two new kinematic-algorythms, on pain, functional disability and kinesiophobia.

Design:

A randomized double blinded placebo controlled trial with double arms in accordance with the CONSORT statement.

Subjects:

Patients with non-specific low back pain will be recruting from Saint-Luc hospital, only a subgroup of them will be included according to specific inclusion criteria tailored for indication of application of SNAG's therapy (Mulligan technique applied on the lumbar spine).

Method:

Subjects will be randomized in 2 groups; real-SNAG and sham-SNAG groups. All patients will be treated during a single session, and real/sham SNAG will be applied from a sitting position with the belt, and in a flexion direction. Two kinematic-algorythms (ROM and Speed) from a validated kinematic spine model will be used and recorded with an opto-electronic device (BTS-Elite). Pain at rest and during flexion, as well as functional disability and kinesiophobia will be recorded by self-reported measures. These outcomes will be blindly evaluated before and after treatment to compare both groups with " Two-Way-ANOVA " statistic with for factors; time and groups.

ELIGIBILITY:
Inclusion Criteria:

* non-specific LBP, mechanical LBP with a pain in flexion direction, the pain in flexion is reduce with the application of SNAG therapy

Exclusion Criteria:

* specific LBP, non-mechanical LBP, the pain is not release in a flexion direction when SNAG is appllied

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Kinematic spine model (Hidalgo et al 2012 Journal of rehabilitation medicine) | Change from baseline until discharge of treatment (same day, single session)
  Use of quantitative variables for ROM and SPEED kinematic (Logit scores index)

SECONDARY OUTCOMES:
Oswestry Disability questionnaire | change from baseline until 2 weeks after treatment
present pain with visual analog scale (VAS) | change from baseline and after treatment the same day (single session)
Tampa scale for kinesiophobia | change from baseline until two weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- READ LAB / Tour Pasteur / Saint-Luc Hospital, Brussels, Belgium

REFERENCES:
- [Background] Hidalgo B, Hall T, Nielens H, Detrembleur C. Intertester agreement and validity of identifying lumbar pain provocative movement patterns using active and passive accessory movement tests. J Manipulative Physiol Ther. 2014 Feb;37(2):105-15. doi: 10.1016/j.jmpt.2013.09.006. Epub 2014 Jan 6. PMID 24401656
- [Background] Hidalgo B, Gobert F, Bragard D, Detrembleur C. Effects of proprioceptive disruption on lumbar spine repositioning error in a trunk forward bending task. J Back Musculoskelet Rehabil. 2013;26(4):381-7. doi: 10.3233/BMR-130396. PMID 23948825
- [Background] Hidalgo B, Gilliaux M, Poncin W, Detrembleur C. Reliability and validity of a kinematic spine model during active trunk movement in healthy subjects and patients with chronic non-specific low back pain. J Rehabil Med. 2012 Sep;44(9):756-63. doi: 10.2340/16501977-1015. PMID 22847223
- [Background] Moutzouri M, Billis E, Strimpakos N, Kottika P, Oldham JA. The effects of the Mulligan Sustained Natural Apophyseal Glide (SNAG) mobilisation in the lumbar flexion range of asymptomatic subjects as measured by the Zebris CMS20 3-D motion analysis system. BMC Musculoskelet Disord. 2008 Oct 1;9:131. doi: 10.1186/1471-2474-9-131. PMID 18828921